CLINICAL TRIAL: NCT03886311
Title: The TNT Protocol: A Phase 2 Study Using Talimogene Laherparepvec,Nivolumab and Trabectedin as First, Second/Third Line Therapy for Advanced Sarcoma, Including Desmoid Tumor and Chordoma
Brief Title: Talimogene Laherparepvec, Nivolumab and Trabectedin for Sarcoma
Acronym: TNT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Oncology Research Center, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOC-1882
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma
Keywords: marine derived alkaloid; PD1 inhibitor; CTLA4 inhibitor
MeSH Terms: conditions — Sarcoma | interventions — talimogene laherparepvec; Nivolumab; Trabectedin; Solutions

STUDY DESIGN:
Intervention Model Description: Forty male and female patients with advanced sarcoma including desmoid tumor and chordoma will be treated with talimogene laherparepvec, nivolumab and trabectedin will be studied and evaluated for progression free survival at month 12.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Talimogene laherparepvec, Nivolumab and Trabectedin (Experimental): This is an open label phase 2 study using known doses of TALIMOGENE LAHERPAREPVEC injected intratumorally, and NIVOLUMAB AND TRABECTEDIN given intravenously.
  A total of 40 previously untreated and treated patients will receive TRABECTEDIN 1.2 mg/m2 CIV over 24 hours q3 weeks, NIVOLUMAB 240 mg IV over 30 min q 2 weeks and TALIMOGENE LAHERPAREPVEC intratumorally q 2 weeks according to tumor size (see Schematic of Study Design and Imlygic product information; www.accessdata.fda.gov). Patients in this study may continue treatment until significant disease progression (see below for criteria for discontinuation of therapy) or unacceptable toxicity occurs up to one year of therapy.
  Interventions: Drug: Talimogene Laherparepvec 100000000 PFU/1 ML Injection Suspension [IMLYGIC]; Drug: Nivolumab IV Soln 100 MG/10ML; Drug: Trabectedin 0.25 MG/1 VIAL Intravenous Powder for Solution

INTERVENTIONS:
Drug: Talimogene Laherparepvec 100000000 PFU/1 ML Injection Suspension [IMLYGIC] — Talimogene laherparepvec, 1Bil is given intratumorally every 2 weeks according to tumor size
  Other Names: TVEC, Imlygic
Drug: Nivolumab IV Soln 100 MG/10ML — NIVOLUMAB 240 mg IV over 30 min q 2 weeks
  Other Names: Opdivo
Drug: Trabectedin 0.25 MG/1 VIAL Intravenous Powder for Solution — TRABECTEDIN 1.2 mg/m2 CIV over 24 hours q3 weeks
  Other Names: Yondelis

SUMMARY:
This is a Phase 2 study using talimogene laherparepvec, nivolumab, and trabectedin as first, second or third line therapy for advanced sarcoma, including desmoid tumor and chordoma.

DETAILED DESCRIPTION:
This is a Phase 2 study using talimogene laherparepvec, nivolumab, and trabectedin as first, second or third line therapy for advanced sarcoma, including desmoid tumor and chordoma. The primary objective is to determine progression-free survival (PFS) at month 12. The secondary objectives are (1) To evaluate the best overall response (BOR) and duration of response (DOR) by RECIST v1.1 via CT scan or MRI at 6,12,18, and 24 weeks post treatment, (2) To determine progression-free survival rate (PFS) at 6 and 9 months, (3) To determine overall survival rate at 6, 9, and 12 months, (4) To determine the incidence of conversion of an unresectable tumor to a resectable tumor, and (5) To evaluate the incidence of adverse events related to TALIMOGENE LAHERPAREPVEC in combination with nivolumab and trabectedin. The exploraratory objective is to correlate response with immune cell trafficking in the tumor microenvironment (TME) of resected tumors.

The primary endpoint is Progression free survival at month 12. The secondary endpoints are: 1) Best overall response (BOR) and duration of response (DOR) by RECIST v1.1 via CT scan or MRI at 6,12,18 and 24 weeks post treatment, 2) PFS rate at 6 and 9 months

• Overall survival rate at 6, 9, and 12 months, 3) Incidence of conversion of an unresectable tumor to a resectable tumor, 4) Incidence of adverse events related to TALIMOGENE LAHERPAREPVEC in combination with nivolumab and trabectedin. The exploratory endpoint is correlation of response with immune cell trafficking in the tumor microenvironment of resected tumors.

Forty male and female subjects > 18 years of age, of any ethnicity, with advanced sarcoma, including desmoid tumor and chordoma will be treated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the inclusion criteria in order to be eligible to participate in the study, as follows:

  * Male or Female ≥ 18 years of age
  * Pathologically confirmed diagnosis of locally advanced unresectable or metastatic sarcoma including desmoid tumor and chordoma
  * Ability to understand the purposes and risks of the study and has signed and dated a written informed consent form approved by the Investigator's IRB/Ethics Committee
  * Willingness to comply with all study procedures and availability for the duration of the study.
  * Previously untreated or treated patient with measurable disease by RECIST v1.1, and at least, one accessible tumor for intratumoral injection of TALIMOGENE LAHERPAREPVEC
  * ECOG performance status ≤ 1
  * Life expectancy of at least 3 months
  * Acceptable liver function: Bilirubin <1.5 times upper limit of normal (ULN; except subjects with Gilbert Syndrome who must have a total bilirubin level < 3.0 ULN); AST (SGOT), ALT (SGPT) and alk phos < 2.5 x ULN (< 5 x ULN if liver metastases present)
  * Acceptable renal function: Creatinine < 1.5 times ULN
  * Acceptable hematologic status: ANC >1500 cells/μL or greater; Platelet count >100,000/μL or greater; Hemoglobin > 9.0 g/dL or greater
  * INR and PT < 1.5 ULN unless taking anti-coagulation, in which case PT, INR and aPTT must be within therapeutic range of intended use of anticoagulants
  * All women of childbearing potential must have a negative urine or serum pregnancy test within 72 hours of enrollment. If urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required; all subjects must agree to use highly effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 5 months for women and 7 months for men after the last dose.

Exclusion Criteria:

* All individuals meeting any of the exclusion criteria at baseline will be excluded from study participation, as follows:

  * Known active central nervous system (CNS) metastases. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids >10 mg/day of prednisone or equivalent. The exception does not include carcinomatosus meningitis which is excluded regardless of clinical stability.
  * History or evidence of active autoimmune disease that requires systemic treatment (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  * Evidence of clinically significant immunosuppression such as the following: - Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease. - concurrent opportunistic infection. - receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to study treatment.
  * Active herpetic skin lesions or prior complications of HSV-1 infection (e.g., herpetic keratitis or encephalitis).
  * Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use.
  * Previous treatment with TALIMOGENE LAHERPAREPVEC or any other oncolytic virus.
  * Received live vaccine within 28 days prior to study treatment.
  * Prior immunosuppressive, chemotherapy, radiotherapy (in which the field encompassed a planned injection site), biological cancer therapy, or major surgery within 28 days prior to study treatment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to study treatment. Adjuvant hormonal therapy is allowed if appropriate for planned study.
  * Prior radiotherapy in which the field does not overlap the injection sites or nonimmunosuppressive targeted therapy within 14 days prior to study treatment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 14 days prior to study treatment
  * Currently receiving treatment with another investigational device or drug study, or < 28 days since ending treatment with another investigational device or drug study(s).
  * Other investigational procedures while participating in this study are excluded.
  * Known to have acute or chronic active hepatitis B infection.
  * Known to have acute or chronic active hepatitis C infection.
  * Known to have human immunodeficiency virus (HIV) infection.
  * History of other malignancy within the past 5 years with the following exceptions:

    * Adequately treated non melanoma skin cancer without evidence of disease at the time of enrollment;
    * Adequately treated cervical carcinoma in situ without evidence of disease at the time of enrollment;
    * Adequately treated breast ductal carcinoma in situ without evidence of disease at the time of enrollment;
    * Prostatic intraepithelial neoplasia without evidence of prostate cancer at the time of enrollment.
  * Subject has known sensitivity to TALIMOGENE LAHERPAREPVEC, NIVOLUMAB or TRABECTEDIN or any of its components to be administered during dosing.
  * Female subject is pregnant or breast-feeding or planning to become pregnant during study treatment and through 3 months after the last dose of TALIMOGENE LAHERPAREPVEC, NIVOLUMAB or TRABECTEDIN.
  * Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of TALIMOGENE LAHERPAREPVEC, NIVOLUMAB or TRABECTEDIN.
  * Sexually active subjects and their partners unwilling to use male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with TALIMOGENE LAHERPAREPVEC.
  * Subjects who are unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or infants under the age of 3 months, during TALIMOGENE LAHERPAREPVEC treatment and through 30 days after the last dose of TALIMOGENE LAHERPAREPVEC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months
  Progression free survival at month 12

SECONDARY OUTCOMES:
Best overall response and duration of response | 12 months
  • Best overall response (BOR) and duration of response (DOR) by RECIST v1.1 via CT scan or MRI at 6,12,18 and 24 weeks post treatment
Progression free survival rate | Nine months
  Prgoression Free Survival rate at 6 and 9 months
)verall survival rate | 12 months
  Overall survival rate at 6, 9, and 12 months
Convesion to resectable tumor | 12 months
  Incidence of conversion of an unresectable tumor to a resectable tumor
Incidence of adverse events | 12 months
  • Incidence of adverse events related to TALIMOGENE LAHERPAREPVEC in combination with nivolumab and trabectedin

CONTACTS AND LOCATIONS:
Overall Officials: Sant P Chawla, MD, Principal Investigator — Sarcoma Oncology Center
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon EM, Sankhala KK, Chawla N, Chawla SP. Trabectedin for Soft Tissue Sarcoma: Current Status and Future Perspectives. Adv Ther. 2016 Jul;33(7):1055-71. doi: 10.1007/s12325-016-0344-3. Epub 2016 May 27. PMID 27234989
- [Result] Chawla SP, Sankhala KK, Ravicz J, Kang G, Liu S, Stumpf N, Leong B, Kim S, Arasheben S, Tseng WW, Gordon EM. Clinical experience with combination chemo-/immunotherapy using trabectedin and nivolumab for advanced soft tissue sarcoma. J Sarcoma Res. 2018; 2(1):1009.